CLINICAL TRIAL: NCT02205853
Title: An Evaluation of a Patient-directed Strategy Compared With a Multi-faceted Strategy to Implement Physical Cancer Rehabilitation Programmes; a Controlled Before and After Study.
Brief Title: Implementation of Physical Cancer Rehabilitation Programmes in a European Healthcare System.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, Rosella Hermens, Dr, Radboud University Medical Center
Allocation: Non-Randomized | Model: Parallel | Purpose: Health Services Research
Other Study IDs: NKI 2010-4854
Record Dates: First submitted 2014-07-21; First posted 2014-07-31 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-08

CONDITIONS: Cancer; Fatigue
Keywords: Oncology Service Hospital; Patient-centred; Exercise; Neoplasms; Rehabilitation; Qualitative Research; Health Plan Implementation; Quality of Health Care; Guidelines; Quality of Life
MeSH Terms: conditions — Neoplasms; Fatigue; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- The patient-directed (PD) strategy (Other): A single-faceted patient-directed (PD) strategy that will embed the change at patient level.
  Interventions: Other: The patient-directed (PD) strategy
- The multi-faceted (MF) strategy (Other): A multi-faceted (MF) strategy that will embed the change at the patient, professional and organizational levels.
  Interventions: Other: The multi-faceted (MF) strategy

INTERVENTIONS:
Other: The patient-directed (PD) strategy — The patient-directed strategy will be designed to embed the success of implementation of PCRPs by influencing the patients.
  Arms: The patient-directed (PD) strategy
Other: The multi-faceted (MF) strategy — The multi-faceted strategy will be designed to embed the success by not only influencing the patients, but also professionals and organizational aspects.
  Arms: The multi-faceted (MF) strategy

SUMMARY:
The aim of this study is to develop and identify the most effective strategy to implement PCRPs into daily care. We want to assess the added value of a multi-faceted strategy compared with a single-faceted patient-directed strategy.

DETAILED DESCRIPTION:
The aim of this study is to develop and identify the most effective strategy to implement PCRPs into daily care. We want to assess the added value of a multi-faceted strategy compared with a single-faceted patient-directed strategy.

We will conduct a clustered controlled before and after study (CBA) in the Netherlands that compares two strategies to implement PCRPs. The patient-directed (PD) strategy (five hospitals) will focus on change at the patient level. The multi-faceted (MF) strategy (five hospitals) will focus on change at the patient, professional and organizational levels. Eligibility criteria are as follows: (A) patients: adults; preferably (history of) cancer in the gastro-intestinal, reproductive and/or urological system; successful primary treatment; and without recurrence/metastases. (B) Healthcare professionals: involved in cancer care.

A stepwise approach will be followed:

Step 1: Analysis of the current implementation of PCRPs and the examination of barriers and facilitators for implementation, via a qualitative study with patients (four focus groups n = 10-12) and their healthcare workers (four focus groups n = 10-12 and individual interviews n = 30-40) and collecting data on adherence to quality indicators (n = 500 patients, 50 per hospital).

Step 2: Selection and development of interventions to create a PD and MF strategy during expert's roundtable discussions, using the knowledge gained in step 1 and a literature search of the effect of strategies for implementing PCRPs.

Step 3: Test and compare both strategies with a clustered CBA (effectiveness, process evaluation and costs), by data extraction from existing registration systems, questionnaires and interviews. For the effectiveness and cost-effectiveness, n = 500 patients, 50 per hospital. For the process evaluation, n=50 patients, 5 per hospital, and n = 40 healthcare professionals, 4 per hospital.

ELIGIBILITY:
Inclusion Criteria:

patients:

* preferably (history of) cancer in the gastro-intestinal, reproductive and/or urological system; successful primary treatment; and without recurrence/metastases.
* Adults
* Diagnosed in one of the participating hospitals
* Able to read and understand Dutch

Healthcare professionals:

• involved in cancer care in one of the participating hospitals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Primary Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
The percentage of screened patients with the screening tool recommended by the Dutch guideline 'Cancer Rehabilitation'. | baseline and at follow-up
  A pre- and post measurement of 'the percentage of screened patients with the screening tool recommended by the Dutch guideline 'Cancer Rehabilitation'' will be done. The differences between the pre- and post measurement will be measured.
The percentage of referrals to PCRPs where needed, according to the Dutch guideline 'Cancer Rehabilitation'. | baseline and at follow-up
  A pre- and post measurement of 'The percentage of referrals to PCRPs where needed, according to the Dutch guideline 'Cancer Rehabilitation'' will be done. The differences between the pre- and post measurement will be measured.

SECONDARY OUTCOMES:
Quality of life | baseline and at follow-up
  A pre- and post measurement of 'QoL' will be done. The differences between the pre- and post measurement will be measured.
Patientempowerment | baseline and at follow-up
  A pre- and post measurement of 'patientempowerment' will be done. The differences between the pre- and post measurement will be measured.
Remaining quality indicators of the Dutch guideline 'Cancer Rehabilitation'. | baseline and at follow-up
  A pre- and post measurement of ' the Remaining quality indicators of the Dutch guideline 'Cancer Rehabilitation'' will be done. The differences between the pre- and post measurement will be measured.

OTHER OUTCOMES:
Process-evaluation | at follow-up
  The experiences and exposure of patients and professionals with the PD- and MF strategy will be evaluated by interviews.
Cost | at follow-up
  incremental costs and incremental cost-effectiveness ratios (ICERs)

CONTACTS AND LOCATIONS:
Overall Officials: C. IJsbrandy, MD, Principal Investigator — Radboud Univeristy Medical Centre Nijmegen; R.P.M.G. Hermens, PhD, Study Chair — Radboud Univeristy Medical Centre Nijmegen
Locations (1):
- Radboud University Nijmegen Medical Center, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Derived] IJsbrandy C, Ottevanger PB, Groen WG, Gerritsen WR, van Harten WH, Hermens RP. Study protocol: an evaluation of the effectiveness, experiences and costs of a patient-directed strategy compared with a multi-faceted strategy to implement physical cancer rehabilitation programmes for cancer survivors in a European healthcare system; a controlled before and after study. Implement Sci. 2015 Sep 7;10:128. doi: 10.1186/s13012-015-0312-3. PMID 26345182